CLINICAL TRIAL: NCT04556383
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate GB004 in Adult Subjects With Mild-to-moderate Active Ulcerative Colitis
Brief Title: A Study With GB004 in Adult Subjects With Active Ulcerative Colitis (UC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to lack of treatment benefit.
Sponsor: GB004, Inc. (Industry)
Responsible Party: Sponsor
Organization: Gossamer Bio Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GB004-2101; 2020-002306-12 (EudraCT Number)
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Ulcerative Colitis
Keywords: Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects, investigators and site personnel, and the Sponsor will be blinded to individual subject treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PCP Placebo (Placebo Comparator): PCP Placebo for oral administration for 36 weeks
  Interventions: Drug: Placebo
- PCP GB004 480 mg QD (Experimental): PCP GB004 480 mg QD for oral administration for 36 weeks
  Interventions: Drug: GB004
- PCP GB004 480 mg BID (Experimental): PCP GB004 480 mg BID for oral administration for 36 weeks
  Interventions: Drug: GB004
- Open-Label Extension (OLE) GB004 480 mg BID (Experimental): OLE GB004 480 mg BID for oral administration for 24 weeks
  Interventions: Drug: GB004

INTERVENTIONS:
Drug: GB004 — oral tablet
  Arms: Open-Label Extension (OLE) GB004 480 mg BID; PCP GB004 480 mg BID; PCP GB004 480 mg QD
Drug: Placebo — oral tablet
  Arms: PCP Placebo

SUMMARY:
A 2-part study, comprising of a 36-week placebo-controlled period (PCP) and a 24-week open-label extension (OLE) period, to assess the efficacy and safety of 2 dose regimens of GB004 when added to background UC therapy of 5-aminosalicylate (5-ASA) with or without systemic steroids.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects aged ≥ 18 years at the time of signing the informed consent form (ICF) prior to initiation of any study specific activities/procedures.
* UC diagnosed at least 3 months prior to first dose of investigational product (IP) on Day 1.
* Currently receiving treatment for UC, on a stable dose for at least 2 weeks prior to flexible sigmoidoscopy or colonoscopy, with oral 5-ASA (eg, mesalamine, sulfasalazine) alone or with one of the following oral treatments:

  1. prednisone ≤ 20 mg/day or equivalent or
  2. beclomethasone ≤ 5 mg/day or
  3. budesonide or budesonide multi-matrix (MMX) of ≤ 9 mg/day

Exclusion Criteria:

* Prior approved biologic therapy used for the treatment of UC.
* Diagnosis of Crohn's disease, indeterminate colitis, or pouchitis, or presence of bacterial or parasitic infection.
* Tofacitinib, oral cyclosporine, sirolimus or mycophenolate mofetil within 8 weeks of Day 1.
* Azathioprine, or 6-mercaptopurine within 1 day of Day 1.

NOTE: Other Inclusion/Exclusion criteria may apply per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (77):
- United States (13):
  - B G Clinical Research, Inc., Encinitas, California
  - Gastro Care Institute, Lancaster, California
  - Texas Digestive Disease Consultants, Baton Rouge, Louisiana
  - Gastroenterology Clinic of Acadiana, Lafayette, Louisiana
  - Delta Research Partners, Monroe, Louisiana
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Freehold Endoscopy Associates, LLC d/b/a/ Endoscopy Center of Monmouth County, Freehold, New Jersey
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Texas Digestive Disease Consultant, Southlake, Texas
  - Washington Gastroenterology, PLLC, Bellevue, Washington
  - Washington Gastroenterology, PLCC, Tacoma, Washington
- Georgia (5):
  - JSC Infectious Diseases, AIDS and Clinical Immunology Research Center, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - LTD Central University Clinic After Academic N. Kipshidze, Tbilisi
  - LTD Coloproctological Center of Georgia, Tbilisi
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center LTD, Tbilisi
- PMSI Republican Clinical Hospital "Timofei Mosneaga", Chisinau, Moldova
- Poland (14):
  - CLINSANTE Clinical Research Center Civil Law Partnership Ewa Galczak-Nowak, Malgorzata Trzaska, Bydgoszcz
  - St. John Paul 2 Municipal Hospital in Elblag, Department of Internal Medicine, Elblag
  - Clinical Research Center of Karkonosze - Lexmedica Limited Liability Company, KCBK - LEXMEDICA, Jelenia Góra
  - Professor K. Gibinski University Clinical Centre of the Medical University of Silesia in Katowice, Katowice
  - "LANDA" Katarzyna Agata Landa, Landa" Specialist Doctor's Offices, Krakow
  - Medicome Limited Liability Company, Oswiecim Clinical Trial Centre, Oświęcim
  - Marek Horynski, MD, Ph.D. Individual Specialist Medical Practice [Specjialistyczna Praktyka Lekarska Dr med. Marek Horynski], Sopot
  - "NOWE ZDROWIE-CK" Kieltucki and Partners General Partnership, NOWE ZDROWIE-CK, Staszów
  - "Gastromed" Torun Gastrology Centre [Torunskie Centrum Gastrologiczne "Gastromed"], Torun
  - EB GROUP Limited Liability Company, MDM Health Centre, Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Reuma Park Clinic Limited Liability Company Limited Partnership, Reuma Park Medical Center, Warsaw
  - VIVAMED Non-Public Healthcare Facility, Warsaw
  - Clinical Research Center Piotr Napora Medical Doctors Professional Partnership, Wroclaw
- Colentina Clinical Hospital, Bucharest, Romania
- Russia (14):
  - Limited Liability Company Joint Venture Diagnostic Center "Biotherm", Barnaul
  - "Myod" Ltd., Bataysk
  - Federal Siberian Research Clinical Center under the Federal Medical Biological Agency, Krasnoyarsk
  - Moscow State-Funded Healthcare Institution City Clinical Hospital n.a. V.M. Buyanov under Moscow Healthcare Department, Moscow
  - Medical Center SibNovoMed, Limited Liability Company, Novosibirsk
  - Novosibirskiy Gastrocenter, LLC, Novosibirsk
  - Institute of Cytology and Genetics, Siberian Branch of the Russian Academy of Sciences, Novosibirsk
  - Medical Diagnostic Center, Limited Liability Company, Orenburg
  - Penza Regional Clinical Hospital named after N.N. Burdenko, Penza
  - Clinic UZI 4D, Limited Liability Company, Pyatigorsk
  - S.M. Kirov Miltiary Medical Academy, Saint Petersburg
  - St. Petersburg State-Funded Healthcare Institution: City Outpatient Care Unit No. 38, Saint Petersburg
  - Consultation and Diagnostics Center and Outpatient Care Unit under the Department of Presidential Affairs, Saint Petersburg
  - Regional State-Funded Healthcare Institution: Novgorod Regional Clinic Hospital, Veliky Novgorod
- Serbia (6):
  - Clinical Hospital Center "Dr Dragisa Misovic Dedinje'' local lab, Belgrade
  - Clinical Hospital Center "Dr Dragisa Misovic Dedinje'', Belgrade
  - Clinical Hospital Center Zemun, Belgrade
  - Zvezdara University Medical Center-local lab, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - General Hospital "Djordje Joanovic", Zrenjanin
- South Korea (3):
  - Inje University Heaundae Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
- Ukraine (20):
  - Communal Nonprofit Enterprise "Cherkasy Regional Hospital of Cherkasy Oblast Council", Cherkasy
  - Regional Communal Noncommercial Enterprise "Chernivtsi Regional Clinical Hospital" Site 9519, Chernivtsi
  - Regional Communal Noncommercial Enterprise "Chernivtsi Regional Clinical Hospital" Site 9527, Chernivtsi
  - Public Non-Profit Enterprise "Regional Clinical Hospital under Ivano-Frankivsk Regional Council", Ivano-Frankivsk
  - PNPE "Prof. O.O. Shalimov City Clinical Hospital #2" under Kharkiv City Council, Kharkiv
  - Public Non-Profit Enterprise under Kharkiv Regional Council "Regional Clinical Hospital", Kharkiv
  - PNPE "Kyiv City Clinical Hospital #18" under the Executive Body of Kyiv City Council, Kyiv
  - Medical Center of the Limited Liability Company "Harmoniia Krasy", Kyiv
  - Medical Center "OK!Clinic+" of the Company with Limited Liability "International Institute of Clinical Research", Kyiv
  - Medical Center of the Limited Liability Company "Medical Center "CONSILIUM MEDICAL", Kyiv
  - Public Non-Profit Enterprise under Kyiv Regional Council "Kyiv Regional Hospital", Kyiv
  - The Municipal Enterprise "Volyn Regional Clinical Hospital" of the Volyn Regional Council, Lutsk
  - Communal Noncommercial Enterprise of Lviv Regional Council "Lviv Regional Clinical Hospital", Lviv
  - Public Non-Profit Enterprise "Odesa Regional Clinical Hospital" under Odesa Regional Council, Odesa
  - Public Enterprise "Poltava M.V. Sklifosovsky Regional Clinical Hospital under Poltava Regional Council", Poltava
  - MNPE "Vinnytsia Regional Clinical Hospital named after M.I. Pirogov Vinnytsia Regional Council", Vinnytsia
  - Communal Non-Commercial Enterprise "Vinnytsia City Clinical Hospital #1, Vinnytsia
  - PNPE "City Hospital of Urgent and Emergency Medical Care under Zaporizhia City Council", Zaporizhia
  - MNPE "Zaporizhia Regional Clinical Hospital" of Zaporizhia Regional Council, Zaporizhia
  - Limited Liability Company "Medibor", Zhytomyr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Danese S, Levesque BG, Feagan BG, Jucov A, Bhandari BR, Pai RK, Taylor Meadows K, Kirby BJ, Bruey JM, Olson A, Osterhout R, Van Biene C, Ford J, Aranda R, Raghupathi K, Sandborn WJ. Randomised clinical trial: a phase 1b study of GB004, an oral HIF-1alpha stabiliser, for treatment of ulcerative colitis. Aliment Pharmacol Ther. 2022 Feb;55(4):401-411. doi: 10.1111/apt.16753. Epub 2022 Jan 10. PMID 35014040

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo-Controlled Period (PCP) Placebo: PCP Placebo for oral administration for 36 weeks
Period: PCP
Arm/Group | Placebo-Controlled Period (PCP) Placebo | PCP GB004 480 mg QD | PCP GB004 480 mg BID | Open-Label Extension (OLE) GB004 480 mg BID
Started | 78 | 78 | 80 | 0
Completed | 23 | 25 | 26 | 0
Not Completed | 55 | 53 | 54 | 0
Not completed — Lack of Efficacy | 28 | 23 | 23 | 0
Not completed — Study terminated by sponsor | 15 | 13 | 16 | 0
Not completed — Withdrawal by Subject | 8 | 6 | 6 | 0
Not completed — Adverse Event | 1 | 7 | 7 | 0
Not completed — Other, Not Specified | 1 | 2 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Site terminated by sponsor | 0 | 1 | 0 | 0
Period: OLE
Arm/Group | Placebo-Controlled Period (PCP) Placebo | PCP GB004 480 mg QD | PCP GB004 480 mg BID | Open-Label Extension (OLE) GB004 480 mg BID
Started | 0 | 0 | 0 | 130
Completed | 0 | 0 | 0 | 39
Not Completed | 0 | 0 | 0 | 91
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 68
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 10
Not completed — Lack of Efficacy | 0 | 0 | 0 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Other, Not Specified | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCP Placebo | PCP GB004 480 mg QD | PCP GB004 480 mg BID | Total
Number analyzed (Participants) | 78 | 78 | 80 | 236
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.1 (14.86) | 44.3 (13.79) | 45.1 (16.76) | 44.8 (15.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 34 | 31 | 102
  Male | 41 | 44 | 49 | 134
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 77 | 74 | 79 | 230
  Race: Asian | 0 | 3 | 0 | 3
  Race: Black or African American | 1 | 0 | 1 | 2
  Race: Other | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 75 | 75 | 80 | 230
  Ethnicity: Hispanic or Latino | 3 | 3 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Remission at PCP Week 12
Description: Clinical remission is defined as a Modified Mayo score ≤ 2, with a rectal bleeding subscore of 0, stool frequency subscore of 0 or 1 (with a ≥ 1 point decrease from baseline), and endoscopic subscore of 0 or 1.
  The Modified Mayo score is an endpoint measure composed of: Stool frequency, Rectal bleeding, and Endoscopic subscores (where the Endoscopic subscore value of 1 does not include friability), each ranging from 0 to 3, that are summed to give a total score ranging from 0 to 9 points, with higher scores indicating greater severity.
Time Frame: At PCP Week 12
Population: PCP Intent to Treat (ITT) Population: all participants who were randomized and received at least 1 dose of PCP study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PCP Placebo | PCP GB004 480 mg QD | PCP GB004 480 mg BID
Number analyzed (Participants) | 78 | 78 | 80
percentage of participants | 17.9 [11.0 to 27.9] | 15.4 [9.0 to 25.0] | 22.5 [14.7 to 32.8]
Statistical Analysis 1: Comparison: PCP Placebo vs PCP GB004 480 mg QD; Test type: Superiority; p = 0.6694, Cochran-Mantel-Haenszel; Risk Difference (RD) = -2.6, 95% CI 2-sided [-15.2 to 10.2] — PCP GB004 480 mg QD vs Placebo
Statistical Analysis 2: Comparison: PCP Placebo vs PCP GB004 480 mg BID; Test type: Superiority; p = 0.4719, Cochran-Mantel-Haenszel; Risk Difference (RD) = 4.6, 95% CI 2-sided [-9.0 to 17.8] — PCP GB004 480 mg BID vs Placebo

2. Primary Outcome: Percentage of Participants With a Treatment Emergent Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a participant, whether or not considered related to study treatment. Abnormal laboratory test results or other safety assessments, including those that worsened from baseline, that were considered clinically significant in the medical and scientific judgment of the investigator were to be reported as AEs. An AE was considered treatment-emergent to the OLE if it started on or after the first dose of OLE study treatment.
Time Frame: From first dose of OLE study treatment through OLE Week 28
Population: OLE Safety Population: all participants who received at least 1 dose of OLE study treatment
Measure: Number; unit: percentage of participants
Groups:
- OLE GB004 480 mg BID: OLE GB004 480 mg BID for oral administration for 24 weeks
Arm/Group | OLE GB004 480 mg BID
Number analyzed (Participants) | 130
percentage of participants | 32.3

3. Secondary Outcome: Percentage of Participants With Clinical Response at PCP Week 12
Description: Clinical response is defined as a reduction in Modified Mayo score of ≥ 2 points and ≥ 35% from baseline, including a decrease in rectal bleeding subscore of ≥ 1 or absolute rectal bleeding subscore of ≤ 1.
  The Modified Mayo score is an endpoint measure composed of: Stool frequency, Rectal bleeding, and Endoscopic subscores (where the Endoscopic subscore value of 1 does not include friability), each ranging from 0 to 3, that are summed to give a total score ranging from 0 to 9 points, with higher scores indicating greater severity.
Time Frame: At PCP Week 12
Population: PCP ITT Population: all participants who were randomized and received at least 1 dose of PCP study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PCP Placebo | PCP GB004 480 mg QD | PCP GB004 480 mg BID
Number analyzed (Participants) | 78 | 78 | 80
percentage of participants | 42.3 [32.0 to 53.4] | 34.6 [25.0 to 45.7] | 52.5 [41.7 to 63.1]
Statistical Analysis 1: Comparison: PCP Placebo vs PCP GB004 480 mg QD; Test type: Superiority; p = 0.3263, Cochran-Mantel-Haenszel; Risk Difference (RD) = -7.7, 95% CI 2-sided [-23.2 to 8.3] — PCP GB004 480 mg QD vs Placebo
Statistical Analysis 2: Comparison: PCP Placebo vs PCP GB004 480 mg BID; Test type: Superiority; p = 0.2002, Cochran-Mantel-Haenszel; Risk Difference (RD) = 10.2, 95% CI 2-sided [-6.1 to 25.8] — PCP GB004 480 mg BID vs Placebo

4. Secondary Outcome: Percentage of Participants With Histologic Remission at PCP Week 12
Description: Histologic remission is defined as Robarts Histopathology Index (RHI) ≤ 3 with lamina propria neutrophils RHI subscore = 0 and neutrophils in epithelium RHI subscore = 0. Histologic remission is evaluated among subjects with both baseline lamina propria neutrophils and neutrophils in epithelium RHI subscores > 0.
  The RHI is a validated instrument that measures histologic disease activity and consists of 4 subscores (chronic inflammatory infiltrate, lamina propria neutrophils, neutrophils in epithelium, and erosion or ulceration). Each subscore ranges from 0-3, with higher subscores indicating greater histologic disease activity. The RHI score is calculated as: (1 x chronic inflammatory infiltrate) + (2 x lamina propria neutrophils) + (3 x neutrophils in epithelium) + (5 x erosion or ulceration). The RHI therefore ranges from 0-33, with higher scores indicating greater histologic disease activity.
Time Frame: At PCP Week 12
Population: Participants in the PCP ITT Population (all participants who were randomized and received at least 1 dose of PCP study treatment) with baseline lamina propria neutrophils and neutrophils in the epithelium RHI subscores > 0.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PCP Placebo | PCP GB004 480 mg QD | PCP GB004 480 mg BID
Number analyzed (Participants) | 69 | 68 | 70
percentage of participants | 26.1 [17.2 to 37.5] | 26.5 [17.4 to 38.0] | 32.9 [23.0 to 44.5]
Statistical Analysis 1: Comparison: PCP Placebo vs PCP GB004 480 mg QD; Test type: Superiority; p = 0.9472, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.4, 95% CI 2-sided [-15.2 to 15.9] — PCP GB004 480 mg QD vs Placebo
Statistical Analysis 2: Comparison: PCP Placebo vs PCP GB004 480 mg BID; Test type: Superiority; p = 0.3685, Cochran-Mantel-Haenszel; Risk Difference (RD) = 6.8, 95% CI 2-sided [-9.3 to 22.4] — PCP GB004 480 mg BID vs Placebo

5. Secondary Outcome: Percentage of Participants With Endoscopic Improvement at PCP Week 12
Description: Endoscopic improvement is defined as an endoscopic subscore of 0 or 1.
  The endoscopic subscore is a component of the Modified Mayo score and is assessed on a 0-3 scale: 0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern); 2 = Moderate disease (marked erythema, absent vascular pattern, friability, erosions); and 3 = Severe disease (spontaneous bleeding, ulceration). Higher scores indicate greater endoscopic disease severity. An endoscopic subscore of 1 does not include friability; an endoscopy with friability is assessed an endoscopic subscore of at least 2.
Time Frame: At PCP Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- PCP GB004 480 m BID: PCP GB004 480 mg BID for oral administration for 36 weeks
Arm/Group | PCP Placebo | PCP GB004 480 mg QD | PCP GB004 480 m BID
Number analyzed (Participants) | 78 | 78 | 80
percentage of participants | 21.8 [14.1 to 32.2] | 23.1 [15.1 to 33.6] | 30.0 [21.1 to 40.8]
Statistical Analysis 1: Comparison: PCP Placebo vs PCP GB004 480 mg QD; Test type: Superiority; p = 0.8484, Cochran-Mantel-Haenszel; Risk Difference (RD) = 1.3, 95% CI 2-sided [-12.7 to 15.2] — PCP GB004 480 mg QD vs Placebo
Statistical Analysis 2: Comparison: PCP Placebo vs PCP GB004 480 m BID; Test type: Superiority; p = 0.2392, Cochran-Mantel-Haenszel; Risk Difference (RD) = 8.2, 95% CI 2-sided [-6.4 to 22.3] — PCP GB004 480 mg BID vs Placebo

6. Secondary Outcome: Percentage of Participants With Mucosal Healing at PCP Week 12
Description: Mucosal healing is defined as endoscopic improvement and histologic remission.
  Please see Secondary Outcome Measure Descriptions above for Percentage of Participants With Endoscopic Improvement at PCP Week 12 and for Percentage of Participants With Histologic Remission at PCP Week 12 for information on the measures of endoscopic improvement and histologic remission, respectively.
Time Frame: At PCP Week 12
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PCP Placebo | PCP GB004 480 mg QD | PCP GB004 480 mg BID
Number analyzed (Participants) | 69 | 68 | 70
percentage of participants | 17.4 [10.2 to 28.0] | 16.2 [9.3 to 26.7] | 20.0 [12.3 to 30.8]
Statistical Analysis 1: Comparison: PCP Placebo vs PCP GB004 480 mg QD; Test type: Superiority; p = 0.8493, Cochran-Mantel-Haenszel; Risk Difference (RD) = -1.2, 95% CI 2-sided [-14.8 to 12.5] — PCP GB004 480 mg QD vs Placebo
Statistical Analysis 2: Comparison: PCP Placebo vs PCP GB004 480 mg BID; Test type: Superiority; p = 0.6647, Cochran-Mantel-Haenszel; Risk Difference (RD) = 2.6, 95% CI 2-sided [-11.5 to 16.5] — PCP GB004 480 mg BID vs Placebo

7. Secondary Outcome: Percentage of Participants With Clinical Remission at PCP Week 36
Description: as for outcome 1
Time Frame: At PCP Week 36
Population: PCP ITT Population: all participants who were randomized and received at least 1 dose of PCP study treatment. Participants who did not consent to protocol version 2.0 and participants who withdrew from PCP due to study termination by Sponsor are excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PCP Placebo | PCP GB004 480 mg QD | PCP GB004 480 mg BID
Number analyzed (Participants) | 63 | 64 | 62
percentage of participants | 14.3 [7.7 to 25.0] | 7.8 [3.4 to 17.0] | 12.9 [6.7 to 23.4]
Statistical Analysis 1: Comparison: PCP Placebo vs PCP GB004 480 mg QD; Test type: Superiority; p = 0.2263, Cochran-Mantel-Haenszel; Risk Difference (RD) = -6.5, 95% CI 2-sided [-19.1 to 6.0] — PCP GB004 480 mg QD vs Placebo
Statistical Analysis 2: Comparison: PCP Placebo vs PCP GB004 480 mg BID; Test type: Superiority; p = 0.8259, Cochran-Mantel-Haenszel; Risk Difference (RD) = -1.4, 95% CI 2-sided [-14.8 to 12.2] — PCP GB004 480 mg BID vs Placebo

8. Secondary Outcome: Percentage of Participants With Clinical Response at PCP Week 36
Description: as for outcome 3
Time Frame: At PCP Week 36
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PCP Placebo | PCP GB004 480 mg QD | PCP GB004 480 mg BID
Number analyzed (Participants) | 63 | 64 | 62
percentage of participants | 20.6 [12.5 to 32.2] | 23.4 [14.7 to 35.1] | 29.0 [19.2 to 41.3]
Statistical Analysis 1: Comparison: PCP Placebo vs PCP GB004 480 mg QD; Test type: Superiority; p = 0.7418, Cochran-Mantel-Haenszel; Risk Difference (RD) = 2.8, 95% CI 2-sided [-12.7 to 18.1] — PCP GB004 480 mg QD vs Placebo
Statistical Analysis 2: Comparison: PCP Placebo vs PCP GB004 480 mg BID; Test type: Superiority; p = 0.2758, Cochran-Mantel-Haenszel; Risk Difference (RD) = 8.4, 95% CI 2-sided [-7.8 to 24.2] — PCP GB004 480 mg BID vs Placebo

9. Secondary Outcome: Percentage of Participants With Histologic Remission at PCP Week 36
Description: Histologic remission is defined as Robarts Histopathology Index (RHI) ≤ 3 with lamina propria neutrophils RHI subscore = 0 and neutrophils in epithelium RHI subscore = 0.
  The RHI is a validated instrument that measures histologic disease activity and consists of 4 subscores (chronic inflammatory infiltrate, lamina propria neutrophils, neutrophils in epithelium, and erosion or ulceration). Each subscore ranges from 0-3, with higher subscores indicating greater histologic disease activity. The RHI score is calculated as: (1 x chronic inflammatory infiltrate) + (2 x lamina propria neutrophils) + (3 x neutrophils in epithelium) + (5 x erosion or ulceration). The RHI therefore ranges from 0-33, with higher scores indicating greater histologic disease activity.
Time Frame: At PCP Week 36
Population: Participants in the PCP ITT Population (all participants who were randomized and received at least 1 dose of PCP study treatment) with baseline lamina propria neutrophils and neutrophils in the epithelium RHI subscores > 0. Participants who did not consent to protocol version 2.0, participants who withdrew from PCP due to study termination by Sponsor, and participants for whom biopsies were collected and not centrally read due to study termination by Sponsor are excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PCP Placebo | PCP GB004 480 mg QD | PCP GB004 480 mg BID
Number analyzed (Participants) | 49 | 48 | 50
percentage of participants | 14.3 [7.1 to 26.7] | 8.3 [3.3 to 19.6] | 16.0 [8.3 to 28.5]
Statistical Analysis 1: Comparison: PCP Placebo vs PCP GB004 480 mg QD; Test type: Superiority; p = 0.3504, Cochran-Mantel-Haenszel; Risk Difference (RD) = -6.0, 95% CI 2-sided [-20.6 to 8.9] — PCP GB004 480 mg QD vs Placebo
Statistical Analysis 2: Comparison: PCP Placebo vs PCP GB004 480 mg BID; Test type: Superiority; p = 0.8009, Cochran-Mantel-Haenszel; Risk Difference (RD) = 1.7, 95% CI 2-sided [-14.2 to 17.5] — PCP GB004 480 mg BID vs Placebo

10. Secondary Outcome: Percentage of Participants With Endoscopic Improvement at PCP Week 36
Description: as for outcome 5
Time Frame: At PCP Week 36
Population: PCP ITT Population: all participants who were randomized and received at least 1 dose of PCP study treatment. Subjects who did not consent to protocol version 2.0 and subjects who withdrew from PCP due to study termination by Sponsor are excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PCP Placebo | PCP GB004 480 mg QD | PCP GB004 480 mg BID
Number analyzed (Participants) | 63 | 64 | 62
percentage of participants | 15.9 [8.9 to 26.8] | 15.6 [8.7 to 26.4] | 12.9 [6.7 to 23.4]
Statistical Analysis 1: Comparison: PCP Placebo vs PCP GB004 480 mg QD; Test type: Superiority; p = 0.9474, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.2, 95% CI 2-sided [-14.3 to 13.7] — PCP GB004 480 mg QD vs Placebo
Statistical Analysis 2: Comparison: PCP Placebo vs PCP GB004 480 mg BID; Test type: Superiority; p = 0.6409, Cochran-Mantel-Haenszel; Risk Difference (RD) = -3.0, 95% CI 2-sided [-16.6 to 10.8] — PCP GB004 480 mg BID vs Placebo

11. Secondary Outcome: Percentage of Participants With Mucosal Healing at PCP Week 36
Description: Mucosal healing is defined as endoscopic improvement and histologic remission.
  Please see Secondary Outcome Measure Descriptions above for Percentage of Participants With Endoscopic Improvement at PCP Week 36 and for Percentage of Participants With Histologic Remission at PCP Week 36 for information on the measures of endoscopic improvement and histologic remission, respectively.
Time Frame: At PCP Week 36
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PCP Placebo | PCP GB004 480 mg QD | PCP GB004 480 mg BID
Number analyzed (Participants) | 49 | 48 | 50
percentage of participants | 14.3 [7.1 to 26.7] | 6.3 [2.1 to 16.8] | 12.0 [5.6 to 23.8]
Statistical Analysis 1: Comparison: PCP Placebo vs PCP GB004 480 mg QD; Test type: Superiority; p = 0.1932, Cochran-Mantel-Haenszel; Risk Difference (RD) = -8.0, 95% CI 2-sided [-22.4 to 6.3] — PCP GB004 480 mg QD vs Placebo
Statistical Analysis 2: Comparison: PCP Placebo vs PCP GB004 480 mg BID; Test type: Superiority; p = 0.7459, Cochran-Mantel-Haenszel; Risk Difference (RD) = -2.3, 95% CI 2-sided [-17.6 to 12.9] — PCP GB004 480 mg BID vs Placebo

ADVERSE EVENTS:
Time Frame: PCP: From first dose in PCP through first dose in OLE (if participant was dosed in OLE) or through PCP Week 40 (if participant was not dosed in OLE) OLE: From first dose in OLE through OLE Week 28
Description: Number of participants at risk based on PCP safety population (all participants who received at least 1 dose of PCP study treatment, grouped according to highest dose of GB004 received) for PCP Reporting Groups and OLE safety population (all participants who received at least 1 dose of OLE study treatment) for OLE Reporting Group. Differences between PCP ITT and safety populations due to 2 participants randomized to GB004 480 mg QD but erroneously received and dosed GB004 480 mg BID.
Arm/Group | PCP Placebo | PCP GB004 480 mg QD | PCP GB004 480 mg BID | OLE GB004 480 mg BID
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/76 | 0/82 | 1/130
Serious Adverse Events (participants affected / at risk) | 2/78 | 2/76 | 4/82 | 9/130
Other Adverse Events (participants affected / at risk) | 13/78 | 29/76 | 27/82 | 8/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCP Placebo (N=78) | PCP GB004 480 mg QD (N=76) | PCP GB004 480 mg BID (N=82) | OLE GB004 480 mg BID (N=130)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 2 | 0 | 4
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PCP Placebo (N=78) | PCP GB004 480 mg QD (N=76) | PCP GB004 480 mg BID (N=82) | OLE GB004 480 mg BID (N=130)
Dizziness (Nervous system disorders) | 1 | 14 | 8 | 0
Nausea (Gastrointestinal disorders) | 2 | 11 | 4 | 0
Somnolence (Nervous system disorders) | 1 | 5 | 7 | 0
Fatigue (General disorders) | 1 | 1 | 5 | 0
Headache (Nervous system disorders) | 0 | 4 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 5 | 0 | 0
COVID-19 (Infections and infestations) | 5 | 4 | 4 | 8
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT04556383/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT04556383/SAP_001.pdf